CLINICAL TRIAL: NCT06415968
Title: Prevalence and Characteristics of Intimate Partner Violence Against Individuals Seeking Hematological Consultations
Acronym: HEMATO-WAST
Status: Terminated | Type: Observational
Why Stopped: difficulty of inclusion, PI decision
Sponsor: Centre Hospitalier Universitaire de Nīmes (Other)
Responsible Party: Sponsor
Other Study IDs: NIMAO/2023-2/JCG-01
Record Dates: First submitted 2024-05-13; First posted 2024-05-16 (Actual); Last update posted 2025-02-18 (Actual); Status verified 2025-02

CONDITIONS: Intimate Partner Violence; Deep Vein Thrombosis (DVT)/Thrombophlebitis; Pulmonary Embolism and Thrombosis
MeSH Terms: conditions — Venous Thrombosis; Pulmonary Embolism; Thrombosis

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Patients presenting at a biological hematology consultation

SUMMARY:
Intimate violence against individuals, which is particularly marked among women, is one of the most widespread human rights violations in the world.

The Women Abuse Screening Tool (WAST) self-questionnaire is a screening tool validated in French.

Our preliminary data describing the association between intimate violence against women and the first attack of unexplained venous thromboembolic disease, show a significant frequency of positive responses to the WAST among women attending a biological hematology consultation at the CHU de Nîmes, for reasons of hemostasis disorders (8% out of the first 200 cases).

The study authors wish to establish the prevalence of this situation among patients presenting to the CHU de Nîmes for hematological exploration and management. They hypothesize that the prevalence of violence against individuals seen in Hematology consultations is higher among individuals with hemostasis pathologies (hemorrhagic and thrombotic pathologies) than those with cellular pathologies, and higher among women than men.

ELIGIBILITY:
Inclusion Criteria:

* Currently in a relationship or has been in one in the last 12 months, regardless of the length of the relationship
* Willing to complete the anonymous WAST self-questionnaire
* able to read and understand French
* Outpatient consultant at Nîmes University Hospital in one of the following departments:

  * Biological hematology consultation
  * Clinical hematology consultation
  * Vascular medicine consultation

Exclusion Criteria:

* Individuals under court protection, guardianship or curatorship
* Individuals unable to read and understand French
* Individuals who have already completed the WAST questionnaire during the study period
* Individuals unable to get away from their partner during the consultation to complete the questionnaire in isolation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Outpatients attending consultations at the CHU de Nîmes for hematological diseases.
Sampling Method: Probability Sample
Enrollment: 138 (Actual)
Dates: Start 2024-09-10 (Actual); Primary Completion 2025-02-11 (Actual); Study Completion 2025-02-11 (Actual)

PRIMARY OUTCOMES:
Prevalence of patients experiencing Intimate Partner Violence according to consulting department | Day 0
  Percentage of patients with a Women Abuse Screening Tool (WAST) score ≥ 5 consulting in the hemostasis pathology versus cellular hematological pathology department. The WAST is an 8-item questionnaire with a score ranging from 0 to 16 (worst violence), with a cut-off of 5 for presence of violence

SECONDARY OUTCOMES:
Prevalence of Intimate Partner Violence in men versus women according to consulting department | Day 0
  WAST score ≥ 5 consulting in the hemostasis pathology versus cellular hematological pathology department in women versus men
Prevalence of Intimate Partner Violence according to patient disease status and gender | Day 0
  WAST questionnaire total score in women versus men, for hemostasis disease versus cellular hematological disease versus hemorrhagic symptomatology versus thrombotic symptomatology
WAST questionnaire score according to patient disease status and gender | Day 0
  Score for individual items of WAST questionnaire in women versus men, for hemostasis disease versus cellular hematological disease versus hemorrhagic symptomatology versus thrombotic symptomatology
Association between the major risk factors for Intimate Partner Violence and WAST score. | Day 0
  WAST questionnaire total score according to: Number of years together, Violence at home growing up, Marital status (divorced or separated), Children living at home, Working status, Finances (personal income, financial difficulties), Living status (together vs separate, size of dwelling, neighbors nearby), Health status of living partner, Health status of patient

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Christophe Gris, Principal Investigator — CHU de Nimes
Locations (1):
- CHU de Nimes, Nîmes, France

IPD SHARING:
Plan to Share IPD: No